CLINICAL TRIAL: NCT04512105
Title: A Phase 1 Open-Label, Dose Escalation Study of Pitavastatin in Combination With Venetoclax in Patients With Chronic Lymphocytic Leukemia or Acute Myeloid Leukemia
Brief Title: Pitavastatin in Combination With Venetoclax for Chronic Lymphocytic Leukemia or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Brem, MD, HS Assistant Clinical Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20205930; CDMRP-CA190644 (Other: Department of Defense); UCI 18-128 (Other: CFCCC)
Record Dates: First submitted 2020-07-03; First posted 2020-08-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; AML, Adult; CLL; CLL, Relapsed; CLL, Refractory
Keywords: Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; AML; CLL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — pitavastatin; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level -1 (DL-1) (Experimental): Patients receive Pitavastatin (PIT) 1 mg PO daily. For CLL patients, they will also receive stabilized Venetoclax (VEN) 400mg PO daily. For AML patients, they will VEN mg PO daily when dosing in combination with azacitidine or decitabine.
  The 1 mg/day dose level will be held in reserve to allow dose reduction in those patients who cannot tolerate DL1.
  Interventions: Drug: Pitavastatin; Drug: Venetoclax
- Dose Level 1 (DL1) (Experimental): Patients receive Pitavastatin (PIT) 2 mg PO daily. For CLL patients, they will also receive stabilized Venetoclax (VEN) 400mg PO daily. For AML patients, they will VEN mg PO daily when dosing in combination with azacitidine or decitabine.
  This is the starting dose level for the study.
  Interventions: Drug: Pitavastatin; Drug: Venetoclax
- Dose Level 2 (DL2) (Experimental): Patients receive Pitavastatin (PIT) 4 mg PO daily. For CLL patients, they will also receive stabilized Venetoclax (VEN) 400mg PO daily. For AML patients, they will VEN mg PO daily when dosing in combination with azacitidine or decitabine.
  If DL1 is well tolerated, the next cohort will progress to this dose level.
  Interventions: Drug: Pitavastatin; Drug: Venetoclax

INTERVENTIONS:
Drug: Pitavastatin — Given PO
  Other Names: LIVALO®
Drug: Venetoclax — Given PO
  Other Names: VENCLEXTA®

SUMMARY:
This is a phase I, dose-escalation, open-label clinical trial determining the safety and tolerability of adding Pitavastatin to Venetoclax in subjects with chronic lymphocytic leukemia (CLL) or acute myeloid leukemia (AML). These are subjects who are newly diagnosed subjects with AML who are ineligible for intensive induction chemotherapy, relapsed/refractory CLL or newly diagnosed CLL.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed AML or CLL, otherwise eligible for VEN-containing therapy at Screening

   1. Newly diagnosed patients with AML deemed ineligible for intensive induction chemotherapy (age 75 and older or < 75 years of age with comorbidities that preclude the use of intensive induction therapy) eligible to receive VEN at Screening. VEN may be combined with azacitidine or decitabine at the discretion of the treating Investigator.
   2. Relapsed/refractory CLL eligible to receive single-agent VEN or VEN in combination with rituximab at Screening.
   3. Newly-diagnosed CLL eligible to receive VEN in combination with obinatuzumab at Screening.
2. Patients who have been receiving stable doses of VEN for at least 5 days prior to initiation of PIT add-on therapy.
3. Age ≥ 18 years.
4. Patients who are already on statins for dyslipidemias are eligible if their previous statin is stopped at least 72 hour prior to starting VEN-based therapy; administration of other statins is prohibited during the study.
5. ECOG performance status ≤ 2 at baseline.
6. Creatinine clearance 30 mL/min or higher; patients assigned to the highest dose level of PIT add-on therapy must have creatinine clearance 60 mL/min or higher.
7. Liver Function tests within the following ranges:

   1. Aspartate aminotransferase (AST) ≤ 3.0 × ULN
   2. Alanine aminotransferase (ALT) ≤ 3.0 × ULN
   3. Bilirubin ≤ 1.5 × ULN (unless elevated bilirubin due to leukemic involvement in the liver or Gilbert's disease)
8. Ability to understand and willingness to sign the informed consent.
9. For the duration of the study treatment period and for at least 90 days following the last dose of study drug female of childbearing potential (FCBP) who are sexually active must agree to employ effective contraceptive methods. Effective contraceptive methods include use of hormonal contraception or an intrauterine device (IUD) by the female partner, or use of condoms by the male partner. An FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
10. For the duration of the study treatment period and for at least 90 days following the last dose of study drug, male patients must agree to use effective contraceptive methods during sexual contact with a female of childbearing potential (FCBP) and must agree to refrain from semen or sperm donation during the same timeframe.

Exclusion Criteria:

1. Patients who are receiving any investigational agents during the previous 30 days or at any time during the study.
2. Patients who have previously received VEN.
3. Patients who satisfy any of the contraindications for PIT.
4. Patients with AML who received prior therapy other than hydroxyurea including those starting hypomethylating therapy for MDS after AML diagnosis.
5. Patients with acute promyelocytic leukemia are excluded
6. Patients with known CNS involvement with leukemia are excluded
7. Patients with active hepatitis B (HBV) or hepatitis C (HCV) infection are excluded. Patients with prior HBV or HCV exposure and those on antiviral medications with negative HBV or HCV viral loads are eligible, as long as the antiretroviral drugs being used do not have significant CYP3A4 interactions.
8. Patients with uncontrolled HIV are excluded. Patients with known HIV and undetectable viral loads are eligible as long as the antiretroviral drugs being used do not have significant CYP3A4 interactions.
9. Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to PEN, PIT, or other statins are excluded.
10. Patients receiving are strong inhibitors or inducers of CYP3A4 within 7 days prior to initiation of VEN therapy are excluded. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. An exception to this is made for patients with AML who require anti-fungal therapy with appropriate dose reduction in VEN (see Section 5.10.2.3).
11. Patients who have consumed grapefruit, grapefruit juice or Seville oranges within 72 hours of initiation of VEN therapy. Consumption of grapefruit, grapefruit juice, Seville oranges, or orange marmalade should be avoided for the duration of the study, as these affect CYP3A4 activity.
12. Patients with certain uncontrolled intercurrent illness are excluded. These include, but are not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illnesses, or social situations that would limit compliance with study requirements.
13. Patients who are pregnant or breastfeeding are excluded.
14. Patients who are unable to swallow pills are excluded.
15. Patients having a malabsorption syndrome or other condition that precludes the oral/enteral route of administration are excluded
16. Patients with an active concurrent malignancy other than CLL or AML are excluded. Patients with a history of definitively treated prior malignancy with low risk of recurrence, skin cancers that have been excised, or on prolonged adjuvant hormonal therapy (ie, for breast or prostate cancer) but are otherwise considered in remission are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose for PIT administered with VEN-containing Standard of Care (SOC) regimens | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  Determination of the maximum tolerated dose (MTD) will be utilized to evaluate the safety and tolerability of adding to PIT to treatment with stable doses of VEN ± anti-CD20 antibodies (patients with CLL) or VEN with hypomethylating agents (patients with AML).
Recommended Phase 2 Dose for PIT administered with VEN-containing SOC regimens | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  Determination of the recommended Phase 2 dose (RP2D) will be utilized to evaluate the safety and tolerability of adding to PIT to treatment with stable doses of VEN ± anti-CD20 antibodies (patients with CLL) or VEN with hypomethylating agents (patients with AML).
Identifying Dose Limiting Toxicities (DLTs) for PIT administered with VEN-containing SOC regimens | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  To evaluate the safety and tolerability of administering PIT in combination with VEN-containing SOC in patients with AML or CLL .
Identifying overall Adverse Event Profile of PIT when given with VEN-containing SOC regimens | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  To evaluate the adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.
Complete Response Rate | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  Primary efficacy endpoint is the complete response rate of subjects who receive PIT when given with VEN-containing SOC regimens. The 2018 International Working Group for Chronic Lymphocytic Leukemia (iwCLL) and 2017 European LeukemiaNet (ELN) definitions of Complete Response (CR) will be utilized to determine the CR rate.

SECONDARY OUTCOMES:
Partial Response Rates | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  Secondary efficacy endpoints are the rates for the other response categories of subjects who receive PIT when given with VEN-containing SOC regimens. The 2018 International Working Group for Chronic Lymphocytic Leukemia (iwCLL) and 2017 European LeukemiaNet (ELN) definitions of Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD) will be utilized to determine the rates for each of these categories.
Stable Disease Rates | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  Secondary efficacy endpoints are the rates for the other response categories of subjects who receive PIT when given with VEN-containing SOC regimens. The 2018 International Working Group for Chronic Lymphocytic Leukemia (iwCLL) and 2017 European LeukemiaNet (ELN) definitions of Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD) will be utilized to determine the rates for each of these categories.
Progressive Disease Rates | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  Secondary efficacy endpoints are the rates for the other response categories of subjects who receive PIT when given with VEN-containing SOC regimens. The 2018 International Working Group for Chronic Lymphocytic Leukemia (iwCLL) and 2017 European LeukemiaNet (ELN) definitions of Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD) will be utilized to determine the rates for each of these categories.
Percentage of Responders | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  Responders are defined as individuals who either received a CR or PR. Responders = CR+PR.
Number of Participants with Abnormal Laboratory Values and/or Adverse Events that Are Related to Treatment | From the start date of treatment until 30 days after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 2 years.
  Changes in safety status, such as Eastern Cooperative Oncology Group (ECOG), performance status, vital signs and laboratory assessments throughout treatment through the trial.

OTHER OUTCOMES:
Composite of PK parameters of VEN and PIT summarized by PIT dose level | Samples will be collected at the following timepoints: Pre-VEN dose during screening, Cycle 1 Day 1 Pre-VEN and PIT dose, Cycle 1 Day 1 Post dose sampling at 1, 2, 4, 8, 24 hours after first PIT dose. Each cycle is 28 days.
  Change in PK parameters from baseline to Cycle 1 to determine if concomitant administration of PIT affects concentrations of VEN when given in combination with PIT.
Composite of dynamic BH3 profiling in priming of ex vivo AML and CLL specimens | Samples will be collected for BH3 profiling at the following timepoints: prior to initiation of VEN treatment, Cycle 1 Day 1 Pre-PIT dose and predose Cycle 1 Day 2. Each cycle is 28 days.
  BH3 profiling on pretreatment and post-treatment bloods samples to assess whether add on treatment with PIT increases apoptotic priming. In dynamic BH3 profiling, the degree of mitochondrial outer membrane permeabilization (MOMP) after exposure to drug is compared to the untreated baseline to quantify the change in priming or induced by exposure to a drug.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Brem, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States